CLINICAL TRIAL: NCT05404243
Title: Randomized Clinical Trial to Test the Efficacy and Safety of Phenolization in Uncomplicated Sacrococcygeal Pilonidal Disease
Brief Title: Clinical Trial to Test the Phenolization in Sacrococcygeal Pilonidal Disease
Acronym: SPQF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HJ23 (Industry)
Responsible Party: Principal Investigator, Jordi Elvira Lopez, Principal investigator, HJ23
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HJ23
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Sacrococcygeal Fistula; Pilonidal Sinus; Pilonidal Disease; Pilonidal Disease of Natal Cleft
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Intervention Model Description: Randomized Clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- phenolization group (Experimental): Curettage of the sacral cyst is performed using a disposable otorhinolaryngologists curette. The perimeter of the cyst is covered with petroleum jelly to protect the skin, and an Abbocath catheter 18 G is introduced into the cystic cavity. Undiluted 88% phenol is instilled into the cavity, ensuring that the cystic cavity is filled. It is maintained for 5 min until complete coagulation of the cyst is achieved.
  Interventions: Drug: phenolization
- conventional surgery (Active Comparator): entire exeresis is performed by means of an electric scalpel
  Interventions: Procedure: Conventional surgery

INTERVENTIONS:
Drug: phenolization — In case of phenolization group, an Abbocath catheter 18 G is introduced into the cystic cavity. Undiluted 88% phenol is instilled into the cavity, ensuring that the cystic cavity is filled. It is maintained for 5 min until complete coagulation of the cyst is achieved.
  Arms: phenolization group
Procedure: Conventional surgery — In case of conventional surgery, entire exeresis is performed by means of an electric scalpel
  Arms: conventional surgery

SUMMARY:
Randomized clinical trial to test the efficacy and safety of phenolization in uncomplicated Sacrococcygeal pilonidal disease

DETAILED DESCRIPTION:
This is a single center randomized controlled clinical trial consisting in 2 treatment groups.

All patients admitted at University Hospital of Tarragona Joan XXIII with Sacrococcygeal pilonidal disease were likely to enter in the study. All patients with uncomplicated sacrococcygeal disease, localized in the midline and with only 1 fistulous orifice.

When the patients met the criteria and after consenting the admission in the study, they were included and were operated. The patients were randomly assigned to the phenolization group or conventional-surgery group. A unique anesthetic and surgical protocol were established for both groups.

Patients in the phenolization group underwent curettage with an otorhinolaryngology spatula and endocavitary phenol with an abocath needle until complete coagulation of the cyst. Patients in the conventional-surgery group were referred to conventional surgery consisting of complete excision of the cyst and closure by second intention. Both groups were managed without admission and discharged within a few hours if they met ALDRETE criteria. They were followed daily by the home hospitalization team

The main endpoint was short or medium-term recurrence of sacrococcygeal disease. The number of recurrences per group and the time from surgery to recurrence were assessed. Secondary endpoints included degree of satisfaction and sick leave

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* ASA (american society anesthesiologists) less than or equal to 3
* patients who live accompanied in a home at a maximum distance of 30 minutes from the hospital
* adequate cognitive capacity

Exclusion Criteria:

* pregnancy or breastfeeding
* complicated Sacrococcygeal pilonidal disease
* non-randomized surgical management

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
recurrence | up to 1 year
  short or medium-term recurrence of sacrococcygeal disease. For this purpose, a clinical follow-up was performed in outpatient clinics where the patient was assessed and explored regularly for signs of recurrence. The number of recurrences per group and the time from surgery to recurrence were assessed

SECONDARY OUTCOMES:
sick leave | up to 1 year
  time from surgery to return to work. This will be counted in days.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordi Elvira Lopez, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No
Only anonymized data on anthropometric characteristics, surgery characteristics, and patient outcomes will be made available.

REFERENCES:
- [Background] Nordon IM, Senapati A, Cripps NP. A prospective randomized controlled trial of simple Bascom's technique versus Bascom's cleft closure for the treatment of chronic pilonidal disease. Am J Surg. 2009 Feb;197(2):189-92. doi: 10.1016/j.amjsurg.2008.01.020. Epub 2008 Jul 17. PMID 18639221
- [Background] Karydakis GE. New approach to the problem of pilonidal sinus. Lancet. 1973 Dec 22;2(7843):1414-5. doi: 10.1016/s0140-6736(73)92803-1. No abstract available. PMID 4128725
- [Background] Bascom J. Pilonidal disease: origin from follicles of hairs and results of follicle removal as treatment. Surgery. 1980 May;87(5):567-72. PMID 7368107
- [Background] Sondenaa K, Andersen E, Nesvik I, Soreide JA. Patient characteristics and symptoms in chronic pilonidal sinus disease. Int J Colorectal Dis. 1995;10(1):39-42. doi: 10.1007/BF00337585. PMID 7745322
- [Background] Dag A, Colak T, Turkmenoglu O, Sozutek A, Gundogdu R. Phenol procedure for pilonidal sinus disease and risk factors for treatment failure. Surgery. 2012 Jan;151(1):113-7. doi: 10.1016/j.surg.2011.07.015. Epub 2011 Oct 6. PMID 21982072
- [Result] Almajid FM, Alabdrabalnabi AA, Almulhim KA. The risk of recurrence of Pilonidal disease after surgical management. Saudi Med J. 2017 Jan;38(1):70-74. doi: 10.15537/smj.2017.1.15892. PMID 28042633
- [Result] GOODALL P. The aetiology and treatment of pilonidal sinus. A review of 163 patients. Br J Surg. 1961 Sep;49:212-8. doi: 10.1002/bjs.18004921421. No abstract available. PMID 13900261
- [Result] Corman ML. Classic articles in colonic and rectal surgery, Pilonidal Sinus. Dis Colon Rectum. 1981 May-Jun;24(4):324-6. No abstract available. PMID 7016481
- [Result] Arslan S, Okur MH, Basuguy E, Aydogdu B, Zeytun H, Cal S, Tegin S, Azizoglu M. Crystallized phenol for treatment of pilonidal sinus disease in children: a comparative clinical study. Pediatr Surg Int. 2021 Jun;37(6):807-813. doi: 10.1007/s00383-020-04798-7. Epub 2021 Apr 15. PMID 33856512
- [Result] Yuksel ME. Pilonidal sinus disease can be treated with crystallized phenol using a simple three-step technique. Acta Dermatovenerol Alp Pannonica Adriat. 2017 Mar;26(1):15-17. doi: 10.15570/actaapa.2017.4. PMID 28352930